CLINICAL TRIAL: NCT07002853
Title: Nature-based Intervention Program for Sustainable Health in Older People Living With Chronic Non-specific Lower Back Pain (PARC Project 2) - A Feasibility Trial
Brief Title: Nature-based Intervention for Chronic Pain in Older People
Acronym: PARC-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); FUQAC (Unknown)
Responsible Party: Principal Investigator, Rubens da Silva, Professor and Director researcher, Université du Québec à Chicoutimi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1991
Record Dates: First submitted 2025-05-24; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Disease; Chronic Pain (Back / Neck); Older Adults (65 Years and Older)
Keywords: Aging; Chronic pain; Non-specific low back pain; Nature-based interventions; Falls; Forest bathing; Shinrin-yoku; Social; Nature connectedness; Functionning; Physical activity; Mindfulness; Meditation; Rehabilitation; Postural control; Strength; Quality of life; Balance
MeSH Terms: conditions — Chronic Disease; Chronic Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nature-based intervention (Experimental): Nature-based intervention group of once a week (2 hours) for 8 weeks
  Interventions: Other: Nature-based Intervention

INTERVENTIONS:
Other: Nature-based Intervention — Combination of activities in nature such as walking, exercises (strengthening, mobility, balance), mindfulness, guided meditation, forest bathing or Shinrin-Yoku, interpretation of nature, gardening and pain education.

SUMMARY:
The goal of this clinical trial is to learn if a nature-based intervention program has positive effects on the physical and psychosocial health in a group of older participants with chronic non-specific lower back pain. The main questions it aims to answer are:

Will the program improve:

* The physical outcomes such as mobility, strength and balance?
* The psychosocial health outcomes?

Participants will:

* Be assessed before and after the program;
* Participate in one session per week of the intervention.

DETAILED DESCRIPTION:
Nonspecific chronic low back pain is defined as persistent pain located between the lower ribs and the gluteal fold, with no identifiable pathoanatomical cause. It is associated with decreased quality of life, mental well-being, increased work absenteeism, and represents a significant economic burden for both individuals and the healthcare system. In the scientific literature, physical activity remains the primary recommended intervention. Recently, nature-based interventions have also been explored as a potential multidisciplinary ally for the management of chronic pain.

The objective of this study is to examine the effects of outdoor physical activity (i.e. walking, general back mobility and strengthening) combined with other nature interventions (i.e. shinrin-yoku, meditation, gardening and pain education) in a group of older adults living with chronic non-specific lower back pain. The intervention will consist of an 8-week group program, conducted once a week for 2 hours. A total of 15 participants will take part in the program to evaluate its impact on both physical and mental health.

Data collection will include both quantitative and qualitative measures. Quantitative outcomes will assess pain disability, quality of life, kinesiophobia (fear of movement), fear of falling, pain catastrophisation, pain beliefs, well-being, depression, nature connectedness, and physical function through standardized tests (e.g., 5 Times Sit to Stand Test), postural control, and gait patterns. Statistical analyses will be performed to compare pre- and post-intervention outcomes, as well as to explore associations between clinical variables, using SPSS software.

Qualitative data will be collected through individual interviews conducted before and at the end of the program to provide a richer understanding of participants' experiences of pain and perceived effects of the program. Interview transcripts will be analyzed using NVivo software.

It is anticipated that this type of intervention will have positive effects for this population and may be considered a promising rehabilitation approach for the management of chronic low back pain in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years +
* Having low back pain for 3 months or more
* Being able to walk independently
* Mental state >25/30 in the MMSE questionnaire
* Frailty score <3/5 (Fried criterias)

Exclusion Criteria:

* Presenting other severe musculoskeletal, cardiovascular, or neurological conditions, or systemic diseases (e.g., cancer).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postural control | change from baseline at 0 to 8 weeks
  Measures of center of pressure (COP) using a force platform during different balance tasks
Trunk postural control on wobble chair | change from baseline at 0 to 8 weeks
  This test measures trunk postural balance during a sitting balance task on an unstable chair where only lumbar spine movements are allowed to restore balance. Briefly, the base of the chair consists of a pivot at its center and four springs that can be arranged and fixed at a distance varying between 6.0 and 21 cm from the center, allowing the system's level of stability to be varied. The system allows only forward/backward and lateral tilting.
Walking | change from baseline at 0 to 8 weeks
  Gait parameters from GaitRite measurement: The participants will be asked to walk at normal and fast speeds on a GaitRite treadmill (GAI-TRite® Platinum Plus System 16' - 4.876 m, SN: Q209, CIR Systems Inc., Franklin, NJ, USA).
  Participants will perform each task twice. Main gait parameters will be used as main outcomes such as velocity in m/s.
Well-being state (WHO-5) | change from baseline at 0 to 8 weeks
  The World Health Organization Well-Being Index (WHO-5) is a widely used self-reported questionnaire designed to measure subjective well-being. It assesses the individual's overall psychological well-being and quality of life. The WHO-5 consists of five simple questions that ask respondents to rate their well-being over the past two weeks. The questions cover aspects such as positive mood, vitality, and general interest in life.The questionnaire is scored on a scale from 0 to 100, with higher scores indicating better well-being.
Depression state (PHQ-9) | change from baseline at 0 to 8 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, monitor, and measure the severity of depression. It consists of nine questions based on the diagnostic criteria for major depressive disorder in the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition).Respondents rate how often they have experienced each symptom over the past two weeks on a scale ranging from 0 (not at all) to 3 (nearly every day). The scores are then added together to produce a total score ranging from 0 to 27, with higher scores indicating greater severity of depressive symptoms
Connection to nature (CNS) | change from baseline at 0 to 8 weeks
  The Connectedness to Nature Scale (CNS) is a psychological assessment tool designed to measure an individual's subjective connection to nature. It evaluates the degree to which people perceive themselves as a part of the natural world and the extent to which they appreciate and value nature in their lives. Respondents are asked to rate their agreement with each statement on a Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The scores are then totaled to provide an overall measure of an individual's connection to nature.
Social Loneliness and Isolation (ÉSUL) | change from baseline at 0 to 8 weeks
  The Échelle de Solitude de l'Université Laval (ÉSUL) is a French-language adaptation of the UCLA Loneliness Scale, developed and validated in Quebec. It is a 20-item self-report questionnaire designed to assess perceived loneliness and social isolation. Each item is rated on a 4-point Likert scale ranging from "Never" to "Often," with higher scores indicating greater feelings of loneliness. The ESUL is commonly used in research and clinical settings involving French-speaking populations.
Interoceptive Awareness (MAIA-Fr) | change from baseline at 0 to 8 weeks
  The Multidimensional Assessment of Interoceptive Awareness - French version (MAIA-Fr) is a validated French-language adaptation of the original MAIA questionnaire. It consists of 32 self-report items grouped into eight subscales that assess different dimensions of interoceptive body awareness, such as Noticing, Emotional Awareness, Self-Regulation, and Body Listening. Items are rated on a 6-point Likert scale ranging from "never" to "always," with higher scores indicating greater interoceptive awareness.
Pain measures | change from baseline at 0 to 8 weeks
  Pain measurement will be done using the Brain pain inventory (BPI) questionnaire. The interference items will be presented with 0-10 scales, with 0=no interference and 10=interferes completely.
Social Provisions (SPS-10) | change from baseline at 8 to 12 weeks
  The Social Provisions Scale-10 (SPS-10) is a shorter version of the original Social Provisions Scale (SPS). It is a brief self-report questionnaire designed to measure perceived social support across five dimensions. The SPS-10 is derived from the longer SPS but consists of a subset of items that capture key aspects of social support.
  Similar to the original SPS, respondents rate their agreement with each item on a Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The SPS-10 provides a quick and efficient way to assess an individual's perceived social support network and their satisfaction with various aspects of their social relationships.
Disability related to low back pain (RMDQ) | change from baseline at 0 to 8 weeks
  The Roland-Morris Disability Questionnaire (RMDQ) is a widely used self-report measure designed to assess physical disability due to low back pain. It consists of 24 yes/no items related to daily physical activities and functional limitations caused by back pain. Each affirmative response scores one point, for a total score ranging from 0 (no disability) to 24 (maximum disability). Higher scores indicate greater functional impairment.
Mood states (POMS-SF) | Before and after each intervention session
  The Profile of Mood States - Short Form (POMS-SF), French Version is a validated self-report questionnaire used to assess short-term changes in mood states. This version consists of 20 items rated on a 5-point Likert scale from 0 ("not at all") to 4 ("extremely"), and measures six mood dimensions: Anxiety (ANX), Depression (DEP), Anger (COL), Vigor (VIG), Fatigue (FAT), and Confusion (CON). Subscale scores are summed separately, with higher scores indicating greater intensity of the respective mood state, except for Vigor, where higher scores reflect better mood. This version, adapted and validated in French by Fillion & Gagnon (1999), is administered before and after each intervention session to assess immediate psychological effects.

SECONDARY OUTCOMES:
Functional mobility test (TUG) | change from baseline at 0 to 8 weeks
  To assess mobility. Equipment: A stopwatch. Directions: Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
5 times Sit-To-Stand (FTSTS) | change from baseline at 0 to 8 weeks
  The Five Times Sit to Stand Test (5xSTS) is a standardized functional assessment used to evaluate lower limb strength, balance, and functional mobility. Participants are instructed to rise from a standard chair and sit back down five times as quickly as possible without using their arms. The total time to complete the five repetitions is recorded in seconds. This measure is commonly used to assess physical function and fall risk in older adults.
Grip strength | change from baseline at 0 to 8 weeks
  Jamar dynamometer to assess maximal isometric hand grip strength and frailty criteria. 3 trials of maximal contraction up 5 seconds. The best value is retained and corrected by body mass index from Fried classification.
Walking speed on 10 metres | change from baseline at 0 to 8 weeks
  Walking speed executed in 10 meter walking test. 2 trials and the best value in time seconds is retained for analysis.
Pain catastrophisation (PCS) | change from baseline at 0 to 8 weeks
  The Pain Catastrophizing Scale (PCS) is a validated self-report questionnaire designed to assess catastrophic thinking related to pain. It consists of 13 items that measure three dimensions: rumination, magnification, and helplessness. Participants rate each item on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("all the time"). The total score ranges from 0 to 52, with higher scores indicating greater levels of pain catastrophizing. The PCS is widely used in both clinical and research settings to evaluate psychological responses to pain.
Kinesiophobia (TSK) | change from baseline at 0 to 8 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a validated self-report questionnaire used to assess fear of movement and re-injury related to physical activity. It consists of 17 items rated on a 4-point Likert scale, ranging from 1 ("strongly disagree") to 4 ("strongly agree"). Total scores range from 17 to 68, with higher scores indicating greater fear of movement. The TSK is commonly used in populations with chronic pain to evaluate the psychological impact of pain on physical activity and rehabilitation outcomes.
Fear and beliefs regarded pain (FABQ) | change from baseline at 0 to 8 weeks
  The Fear and Beliefs Questionnaire (FBQ) is a self-administered questionnaire designed to assess fear-avoidance beliefs and perceptions related to low back pain. It evaluates how individuals perceive the harmfulness of movement and physical activity, and how these beliefs may influence their behavior and functional limitations. The FBQ includes items rated on a Likert scale, with higher scores reflecting stronger fear-avoidance beliefs. It is commonly used in clinical and research settings to better understand the psychosocial factors contributing to chronic pain and disability.

OTHER OUTCOMES:
Falls Efficacy Scale-International (FES-I) | change from baseline at 0 to 8 weeks
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity. The level of concern is measured on a four point Likert scale (1=not at all concerned to 4=very concerned)
Cognitive status | Only at baseline from Sample characterization
  Mini-mental state questionnaire (MMSE or Folstein), which is used for grading the cognitive state of patients in this study. It's assessing the attention and orientation, memory, registration, recall, calculation, language and ability to draw a complex polygon. It is ranged from 0 to 30, where 30 means no impairment.
Frailty criteria from Fried | Only at baseline from Sample characterization
  The presence of frailty criteria according to Fried was assessed with self-report questions and two physical tests from five characteristics : 1) Low physical activity (to capture history of sedentary behavior or activity: ex. Do you get any physical exercise for the sake of exercising? How often do you leave your house?); 2) fatigue (complaint of exhaustion with normal activity such as walking outside, climbing stairs: ex. I felt that everything I did was an effort in the last week?); 3) weight loss (unintentional weight loss 10 lbs. or more in past year or more than 5% in past year); 4) weakness (grip strength evaluated with manual dynamometer; in average <30 kg for men and <18 kg for women, but data is normalized by body mass index); 5) slowness or slow walking speed (usual gait speed over 4.57 meters (15 feet); ex. >6.5 seconds, dependent of height).

CONTACTS AND LOCATIONS:
Overall Officials: Rubens A. da Silva, Ph.D., Study Director — Université du Québec à Chicoutimi; Marie-Ève Langelier, MD, Study Chair — Université du Québec à Chicoutimi; Émilie Fortin, M.Sc, Principal Investigator — Université du Québec à Chicoutimi; Guillaume Léonard, Ph.D., Study Chair — Université de Sherbrooke
Locations (1):
- Université du Québec à Chicoutimi, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suh JH, Kim H, Jung GP, Ko JY, Ryu JS. The effect of lumbar stabilization and walking exercises on chronic low back pain: A randomized controlled trial. Medicine (Baltimore). 2019 Jun;98(26):e16173. doi: 10.1097/MD.0000000000016173. PMID 31261549
- [Background] Hayden JA, Ellis J, Ogilvie R, Malmivaara A, van Tulder MW. Exercise therapy for chronic low back pain. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD009790. doi: 10.1002/14651858.CD009790.pub2. PMID 34580864
- [Background] Fernandez-Rodriguez R, Alvarez-Bueno C, Cavero-Redondo I, Torres-Costoso A, Pozuelo-Carrascosa DP, Reina-Gutierrez S, Pascual-Morena C, Martinez-Vizcaino V. Best Exercise Options for Reducing Pain and Disability in Adults With Chronic Low Back Pain: Pilates, Strength, Core-Based, and Mind-Body. A Network Meta-analysis. J Orthop Sports Phys Ther. 2022 Aug;52(8):505-521. doi: 10.2519/jospt.2022.10671. Epub 2022 Jun 19. PMID 35722759
- [Background] Dagenais S, Tricco AC, Haldeman S. Synthesis of recommendations for the assessment and management of low back pain from recent clinical practice guidelines. Spine J. 2010 Jun;10(6):514-29. doi: 10.1016/j.spinee.2010.03.032. PMID 20494814
- [Background] Brumitt J, Matheson JW, Meira EP. Core stabilization exercise prescription, part I: current concepts in assessment and intervention. Sports Health. 2013 Nov;5(6):504-9. doi: 10.1177/1941738113502451. PMID 24427424
- [Background] Han JW, Choi H, Jeon YH, Yoon CH, Woo JM, Kim W. The Effects of Forest Therapy on Coping with Chronic Widespread Pain: Physiological and Psychological Differences between Participants in a Forest Therapy Program and a Control Group. Int J Environ Res Public Health. 2016 Feb 24;13(3):255. doi: 10.3390/ijerph13030255. PMID 26927141
- [Background] Li Q, Morimoto K, Kobayashi M, Inagaki H, Katsumata M, Hirata Y, Hirata K, Shimizu T, Li YJ, Wakayama Y, Kawada T, Ohira T, Takayama N, Kagawa T, Miyazaki Y. A forest bathing trip increases human natural killer activity and expression of anti-cancer proteins in female subjects. J Biol Regul Homeost Agents. 2008 Jan-Mar;22(1):45-55. PMID 18394317
- [Background] Li Q. Effects of forest environment (Shinrin-yoku/Forest bathing) on health promotion and disease prevention -the Establishment of "Forest Medicine". Environ Health Prev Med. 2022;27:43. doi: 10.1265/ehpm.22-00160. PMID 36328581
- [Background] Irvine KN, Fisher D, Currie M, Colley K, Warber SL. A Nature-Based Intervention for Promoting Physical Activity in Older Adults: A Qualitative Study Using the COM-B Model. Int J Environ Res Public Health. 2024 Jun 27;21(7):843. doi: 10.3390/ijerph21070843. PMID 39063420
- [Background] Frumkin H, Bratman GN, Breslow SJ, Cochran B, Kahn PH Jr, Lawler JJ, Levin PS, Tandon PS, Varanasi U, Wolf KL, Wood SA. Nature Contact and Human Health: A Research Agenda. Environ Health Perspect. 2017 Jul 31;125(7):075001. doi: 10.1289/EHP1663. PMID 28796634
- [Background] Zhang SK, Gu ML, Zhang T, Xu H, Mao SJ, Zhou WS. Effects of exercise therapy on disability, mobility, and quality of life in the elderly with chronic low back pain: a systematic review and meta-analysis of randomized controlled trials. J Orthop Surg Res. 2023 Jul 19;18(1):513. doi: 10.1186/s13018-023-03988-y. PMID 37468931
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Vlaeyen JWS, Maher CG, Wiech K, Van Zundert J, Meloto CB, Diatchenko L, Battie MC, Goossens M, Koes B, Linton SJ. Low back pain. Nat Rev Dis Primers. 2018 Dec 13;4(1):52. doi: 10.1038/s41572-018-0052-1. PMID 30546064
- [Background] Dionne CE, Dunn KM, Croft PR. Does back pain prevalence really decrease with increasing age? A systematic review. Age Ageing. 2006 May;35(3):229-34. doi: 10.1093/ageing/afj055. Epub 2006 Mar 17. PMID 16547119
- [Background] da Silva RA, Vieira ER, Carvalho CE, Oliveira MR, Amorim CF, Neto EN. Age-related differences on low back pain and postural control during one-leg stance: a case-control study. Eur Spine J. 2016 Apr;25(4):1251-7. doi: 10.1007/s00586-015-4255-9. Epub 2015 Oct 1. PMID 26428907
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Result] Lee I, Choi H, Bang KS, Kim S, Song M, Lee B. Effects of Forest Therapy on Depressive Symptoms among Adults: A Systematic Review. Int J Environ Res Public Health. 2017 Mar 20;14(3):321. doi: 10.3390/ijerph14030321. PMID 28335541
- [Result] Berman MG, Jonides J, Kaplan S. The cognitive benefits of interacting with nature. Psychol Sci. 2008 Dec;19(12):1207-12. doi: 10.1111/j.1467-9280.2008.02225.x. PMID 19121124
- [Result] Vanti C, Andreatta S, Borghi S, Guccione AA, Pillastrini P, Bertozzi L. The effectiveness of walking versus exercise on pain and function in chronic low back pain: a systematic review and meta-analysis of randomized trials. Disabil Rehabil. 2019 Mar;41(6):622-632. doi: 10.1080/09638288.2017.1410730. Epub 2017 Dec 5. PMID 29207885
- [Result] White MP, Alcock I, Grellier J, Wheeler BW, Hartig T, Warber SL, Bone A, Depledge MH, Fleming LE. Spending at least 120 minutes a week in nature is associated with good health and wellbeing. Sci Rep. 2019 Jun 13;9(1):7730. doi: 10.1038/s41598-019-44097-3. PMID 31197192
- [Result] Simone C. Gafner A-VB. Test de 10 mètres de marche 10-Meter Walking Test Kinésithérapie, la Revue. 2022;22(248-249):46-9.
- [Result] Bohannon RW. Reference values for the five-repetition sit-to-stand test: a descriptive meta-analysis of data from elders. Percept Mot Skills. 2006 Aug;103(1):215-22. doi: 10.2466/pms.103.1.215-222. PMID 17037663
- [Result] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Result] Sullivan MJL, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment. 1995;7(4):524-32.
- [Result] French DJ, Roach PJ, Mayes S. Peur du mouvement chez des accidentes du travail: l'Echelle de Kinesiophobie de Tampa (EKT). CANADIAN JOURNAL OF BEHAVIOURAL SCIENCE. 2002;34:28-33.
- [Result] Steigen AM, Bergh D. The Social Provisions Scale: psychometric properties of the SPS-10 among participants in nature-based services. Disabil Rehabil. 2019 Jul;41(14):1690-1698. doi: 10.1080/09638288.2018.1434689. Epub 2018 Feb 5. PMID 29402143
- [Result] Orpana HM, Lang JJ, Yurkowski K. Validation of a brief version of the Social Provisions Scale using Canadian national survey data. Health Promot Chronic Dis Prev Can. 2019 Dec;39(12):323-332. doi: 10.24095/hpcdp.39.12.02. PMID 31825785
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Result] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- See also: PARC project 1 for Parkinson Disease — https://www.youtube.com/watch?v=mJKVBMl0Qkk